CLINICAL TRIAL: NCT01293097
Title: Intensive Statin Treatment in Chinese Coronary Artery Disease Patients Undergoing Percutaneous Coronary Intervention(PCI)
Brief Title: Intensive Statin Treatment in Chinese Coronary Artery Disease Patients Undergoing PCI
Acronym: ISCAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of cardiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISCAP
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Non-ST Segment Elevation Myocardial Infarction; Unstable Angina Pectoris; Stable Angina Pectoris
MeSH Terms: conditions — Angina, Unstable; Angina, Stable | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Pravastatin; Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive statin therapy (Active Comparator): Atorvastatin 80mg/d ×2d before PCI. After PCI, atorvastatin 40mg/d until 30 days later, and then followed by usual care
  Interventions: Drug: Atorvastatin
- Usual care (Other): Usual care, but statin dose should not be higher than that described in exclusion criteria.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg/d ×2d before PCI. After PCI, atorvastatin 40mg/d until 30 days later, and then followed by usual care
  Other Names: Liptor
  Arms: Intensive statin therapy
Drug: Statin — Usual care, but statin dose should not be higher than that described in exclusion criteria
  Other Names: Liptor; Zocor; Pravachol; Lescol
  Arms: Usual care

SUMMARY:
This randomized, open label, controlled, parallel group study is designed to test whether 2-day high dose atorvastatin administration before PCI and 30-day continuous intensive atorvastatin treatment is superior to usual care, in terms of peri-PCI cardiovascular events, as well as 6-month prognosis. The goal is to set up an optimized protocol for peri-PCI statin treatment in Chinese CHD patients. Safety will also be observed.

DETAILED DESCRIPTION:
The study objective is to test whether 2-day high dose atorvastatin administration before PCI and 30-day continuous intensive atorvastatin treatment is superior to usual care, in terms of peri-PCI cardiovascular events, as well as 6-month prognosis.

2160 patients with non-ST segment elevated acute coronary syndrome (ACS)or stable angina pectoris (SAP) scheduled for selective PCI are randomized into two groups. The study group is given atorvastatin 80 mg/d×2d before PCI while the control group receives usual care. After angiography, patients who are not undergoing PCI procedure will be excluded from the study as selection failure. After PCI procedure, the study group is given atorvastatin 40mg/d until 30 days after PCI while the control group receive usual care. The last visit will be at 6 months after PCI. Patients data such as troponin, CK-MB, Scr, CCR, ALT, AST before and after procedure will be recorded. 1100 effective patients will be finally enrolled.

The study will be conducted at about 54 centers in China. Data will be collected on 2,100 NSTE or SAP patients undergoing PCI.

Primary outcome: MACE within 30 days after PCI. Secondary outcome: Post-procedural change of inflammatory biomarkers (hs-CRP); Morbidity of CIN; Proportion of patients who experience at least once AST > 3ULN，ALT > 3ULN or CK > 5ULN after initiation of study treatment. Proportion of patients who experience at least once AST, ALT, or CK>ULN after initiation of study treatment; Proportion of patients who take reduced dose of atorvastatin, withdraw study treatment, or withdraw study due to adverse events; Combined endpoint of death, cardiac death, myocardial infarction, heart failure, cardiac hospitalization, revascularization, and cerebrovascular events within 6 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years old
* Patients with clinical diagnosis of NSTE-ACS (unstable angina or NSTE acute myocardial infarction) or stable angina pectoris (SAP) scheduled for selective coronary angiography
* Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Patients presenting with ST-segment elevation acute myocardial infarction (STEMI) or high risk NSTE-ACS, warranting emergency coronary angiography:
* Experienced STEMI within previous 30 days
* Taking or, needing to take atorvastatin over than 20mg/d or any other equivalent statin (such as simvastatin 20mg/d, pravastatin 40mg/d, fluvastatin 80mg/d or rosuvastatin 5mg/d ) in the next 6 months, or needing to take fibrates simultaneously according to investigators' judgment.
* Anticipated repeated PCI within 6 months
* LDL-C < 1.8mmol/L in patients without statin therapy in 1 months
* Endstage congestive heart failure, or LVEF < 30%
* Active hepatic disease or hepatic dysfunction, or AST/ALT > 1.5UNL
* Myopathy or increased creatine kinase (CK>2 UNL)
* White blood cell < 4×109/L or platelet < 100×109/L
* Severe renal dysfunction(Scr > 3 mg/dl or 264μmol/L)
* Allergic or experienced serious adverse reaction to HMG-CoA reductase, or ineligible to take statin as investigator's judgment
* Severe aortic valve stenosis or severe mitral stenosis, Obstructive hypertrophic cardiomyopathy, pericardial diseases
* Pregnancy, lactation, or child bearing potential women without any effective contraception
* Accompanied with malignant disease or other disease, which cause life expectancy < 6 months
* Participating in other interventional clinical trails using drugs or devices
* Patients with any condition which, in the investigator's judgment, might increase the risk to the subject for any adverse event or abnormal laboratory finding

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2884 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
30-day MACEs after PCI | 30 days after PCI
  30-day major adverse cardiovascular events (combined endpoints of cardiac death, myocardial infarction, and target vessel revascularization ) after PCI

SECONDARY OUTCOMES:
Post-procedural change of inflammatory biomarkers (hs-CRP) | 24 hours after PCI
  Post-procedural change of inflammatory biomarkers (hs-CRP)
Morbidity of CIN | 48 hours after PCI
  Morbidity of CIN
Elevation of ALT, AST and CK | 6 months after PCI
  Proportion of patients who experience at least once AST>3UNL，ALT>3UNL or CK>5UNL after initiation of study treatment. Proportion of patients who experience at least once AST, ALT, or CK>UNL after initiation of study treatment.
Adverse events | 6 months after PCI
  Proportion of patients who take reduced dose of atorvastatin, withdraw study treatment, or withdraw study due to adverse events
Combined endpoint of MACEs, cardiac hospitalization and cerebrovascular events | 6 months after PCI
  Combined endpoint of death, cardiac death, myocardial infarction, heart failure, cardiac hospitalization, revascularization, and cerebrovascular events within 6 months after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Division of Cardiology, Peking University First Hospital, Beijing, China